CLINICAL TRIAL: NCT03757156
Title: Aspirin Withdrawal and Clinical Outcome in Patients With Moderate to High Cardiovascular Risk But Without Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2018-0910
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Healthy Participants With Moderate and High Cardiovascular Risk

STUDY DESIGN:
Intervention Model Description: Aspirin maintenance group versus aspirin interruption group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin maintenance group (No Intervention): People who are taking aspirin continue to take aspirin.
- Aspirin withdrawal group (Experimental): People who are taking aspirin stop to taking aspirin.
  Interventions: Other: Withdrawal of aspirin

INTERVENTIONS:
Other: Withdrawal of aspirin — People who are taking aspirin stop to taking aspirin.
  Arms: Aspirin withdrawal group

SUMMARY:
While the efficacy of aspirin for the secondary prevention of cardiovascular disease is evident, the effect of aspirin for primary prevention is unclear. The use of aspirin reduces cardiovascular mortality and myocardial infarction but increases side effects such as bleeding. Therefore, the use of aspirin for primary prevention in people without cardiovascular disease should be determined by individual risk and clinical benefit. The European guidelines have been changed to not recommend aspirin use in people without cardiovascular disease, but there are still people taking aspirin for primary prevention. The purpose of this study is to investigate the effect of aspirin withdrawal on cardiovascular events in patients without cardiovascular disease.

This is a single center, prospective, randomized clinical study evaluating the safety and efficacy of withdrawal of aspirin among patients with moderate or high cardiovascular risk.

DETAILED DESCRIPTION:
Patients taking aspirin will be randomly assigned to a group that maintains taking aspirin and a group that discontinues to take aspirin by 1:1 manner. The follow-up duration is five years and clinical outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-80 years old
* Subjects who are taking for more than 12 months
* Subjects with moderate or high cardiovascular risk based on cardiovascular risk classification of 2015 Korea Society of Lipidology And Atherosclerosis guideline or 2004 American Heart Association guideline: 1) moderate risk: people with ≥2 major risk factors, 2) high risk: people with carotid atherosclerosis, abdominal aortic aneurysm, or diabetes, who is taking statin
* Subjects who voluntarily participate in the study and sign informed consent form

Exclusion Criteria:

* Subjects with a history of major cardiovascular disease confirmed by medical history and medical history; myocardial infarction, angina pectoris, coronary angioplasty, coronary artery bypass surgery, peripheral vascular disease, ischemic stroke, transient ischemic attack
* Subjects has any contraindication to use of aspirin or hypersensitivity to aspirin
* Subjects with atrial fibrillation
* Subjects who are taking anti-platelet agents other than aspirin or anticoagulants
* Subjects who have been diagnosed with cancer within the last 5 years
* Pregnant women or those who have pregnancy plan after enrolling in this study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4118 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events(MACE) | 5 years
  Major adverse cardiovascular events is composite endpoint. It includes cardiovascular death, nonfatal myocardial infarction, nonfatal ischemic stroke, coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft), nonfatal ischemic stroke, and transient ischemic attack.

SECONDARY OUTCOMES:
cardiovascular death | 5 years
  Individual component of primary endpoint
nonfatal myocardial infarction | 5 years
  Individual component of primary endpoint
nonfatal ischemic stroke | 5 years
  Individual component of primary endpoint
coronary revascularization | 5 years
  Individual component of primary endpoint
transient ischemic attack | 5 years
  Individual component of primary endpoint
Bleeding | 5 years
  Major bleeding is defined with International Society on Thrombosis and Haemostasis (ISTH) criteria: 1) fatal bleeding; 2)Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; 3) bleeding causing a fall in hemoglobin level of 2 g/dL or more, or leading to transfuction of two or more units of whole blood or red cells. Bleeding that is not classified as major bleeding is minor.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Cardiovascular Center, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214
- [Background] Bibbins-Domingo K; U.S. Preventive Services Task Force. Aspirin Use for the Primary Prevention of Cardiovascular Disease and Colorectal Cancer: U.S. Preventive Services Task Force Recommendation Statement. Ann Intern Med. 2016 Jun 21;164(12):836-45. doi: 10.7326/M16-0577. Epub 2016 Apr 12. PMID 27064677
- [Background] Saito Y, Okada S, Ogawa H, Soejima H, Sakuma M, Nakayama M, Doi N, Jinnouchi H, Waki M, Masuda I, Morimoto T; JPAD Trial Investigators. Low-Dose Aspirin for Primary Prevention of Cardiovascular Events in Patients With Type 2 Diabetes Mellitus: 10-Year Follow-Up of a Randomized Controlled Trial. Circulation. 2017 Feb 14;135(7):659-670. doi: 10.1161/CIRCULATIONAHA.116.025760. Epub 2016 Nov 15. PMID 27881565
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Wilson PW, D'Agostino RB, Levy D, Belanger AM, Silbershatz H, Kannel WB. Prediction of coronary heart disease using risk factor categories. Circulation. 1998 May 12;97(18):1837-47. doi: 10.1161/01.cir.97.18.1837. PMID 9603539
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Ikeda Y, Shimada K, Teramoto T, Uchiyama S, Yamazaki T, Oikawa S, Sugawara M, Ando K, Murata M, Yokoyama K, Ishizuka N. Low-dose aspirin for primary prevention of cardiovascular events in Japanese patients 60 years or older with atherosclerotic risk factors: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2510-20. doi: 10.1001/jama.2014.15690. PMID 25401325